CLINICAL TRIAL: NCT00001034
Title: A Randomized, Comparative, Placebo-Controlled Trial of the Safety and Efficacy of Oral Ganciclovir for Prophylaxis of Cytomegalovirus (CMV) Retinal and Gastrointestinal Mucosal Disease in HIV-Infected Individuals With Severe Immunosuppression
Brief Title: The Safety and Effectiveness of Ganciclovir in the Prevention of Cytomegalovirus (CMV) of the Eyes and Disease of the Stomach and Intestines in Patients With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 023; 11573 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections; Gastrointestinal Diseases
Keywords: Retinitis; Ganciclovir; Cytomegalovirus Infections; Administration, Oral; Acquired Immunodeficiency Syndrome; Gastrointestinal System
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Gastrointestinal Diseases; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To evaluate the safety and efficacy of oral ganciclovir for prophylaxis against cytomegalovirus (CMV) retinal and gastrointestinal mucosal disease in HIV-infected patients with severe immunosuppression.

The most recent treatments against CMV disease have been ganciclovir and foscarnet. Until recently, both drugs required intravenous administration. An oral form of ganciclovir, if shown to be effective therapy against CMV, would be a more suitable method of administration for prophylaxis.

DETAILED DESCRIPTION:
The most recent treatments against CMV disease have been ganciclovir and foscarnet. Until recently, both drugs required intravenous administration. An oral form of ganciclovir, if shown to be effective therapy against CMV, would be a more suitable method of administration for prophylaxis.

Patients are randomized in a 2:1 ratio to receive either oral ganciclovir or placebo for a minimum of 12 months. PER AMENDMENT 9/19/94: Patients who have not reached a study endpoint may choose to continue blinded prophylaxis or discontinue blinded prophylaxis and begin open-label ganciclovir. PER AMENDMENT 5/2/95: After the common closing date (6/3/95) patients who have not met a CMV end point or experienced a serious toxicity that required permanent discontinuation of active oral ganciclovir will be eligible to receive open-label oral ganciclovir through an open-label extension phase of study 023 until 8/31/95.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Anti-PCP prophylaxis.
* Maintenance or prophylaxis therapy for other opportunistic infections besides CMV.

Patients must have:

* Working diagnosis of HIV infection.
* CD4 count <= 100 cells/mm3.
* Positive CMV serology (IgG) or CMV culture, in the absence of active disease, documented at any time prior to study entry.
* Reasonably good health.
* Life expectancy of at least 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Acute life-threatening illness.
* Active lymphoma.
* Hypersensitivity to acyclovir.
* Lack of willingness or ability, in the opinion of the clinician, to comply with protocol requirements.

Concurrent Medication:

Excluded:

* Vidarabine.
* Amantadine hydrochloride (Symmetrel).
* CMV hyperimmune globulin/intravenous immune globulin.
* Cytarabine.
* Fiacitabine (FIAC) or fialuridine (FIAU).
* Foscarnet.
* Intravenous ganciclovir.
* HPMPC.
* Idoxuridine.
* Intravenous acyclovir.
* Oral acyclovir at > 1 g/day.
* Other drugs with potential anti-CMV activity.

Prior Medication:

Excluded within 60 days prior to study entry:

* Foscarnet.

Excluded within 2 weeks prior to study entry:

* Vidarabine.
* Amantadine hydrochloride (Symmetrel).
* CMV hyperimmune globulin/intravenous immune globulin.
* Cytarabine.
* Fiacitabine (FIAC) or fialuridine (FIAU).
* Ganciclovir.
* HPMPC.
* Idoxuridine.
* Intravenous acyclovir.
* Oral acyclovir at > 1 g/day.
* Other drugs with potential anti-CMV activity.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 850
Dates: Study Completion 1995-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brosgart C, Study Chair; Craig C, Study Chair
Locations (17):
- United States (17):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Schering - Plough Corp, Kenilworth, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Brosgart C, Craig C, Louis TA, Hillman D, Costanzo L, Timpone J, Scott J, Nunley F, Stempien MJ. Design and demographics in a multicenter trial of cytomegalovirus (CMV) prophylaxis in advanced HIV disease. Int Conf AIDS. 1994 Aug 7-12;10(2):10 (abstract no 331B)
- [Background] Brosgart CL, Louis TA, Hillman DW, Craig CP, Alston B, Fisher E, Abrams DI, Luskin-Hawk RL, Sampson JH, Ward DJ, Thompson MA, Torres RA. A randomized, placebo-controlled trial of the safety and efficacy of oral ganciclovir for prophylaxis of cytomegalovirus disease in HIV-infected individuals. Terry Beirn Community Programs for Clinical Research on AIDS. AIDS. 1998 Feb 12;12(3):269-77. doi: 10.1097/00002030-199803000-00004. PMID 9517989